CLINICAL TRIAL: NCT06851741
Title: Behavioural Activation for Depression in Adults with Severe Learning Disabilities. a Feasibility Randomised Controlled Study of Behavioural Activation with Treatment As Usual (TAU) Vs TAU Alone
Brief Title: Behavioural Activation and Severe Learning Disabilities
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GN22MH146
Record Dates: First submitted 2025-02-10; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-11

CONDITIONS: Intellectual Disabilities; Depression
Keywords: Intellectual disability; Depression
MeSH Terms: conditions — Intellectual Disability; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The research assistants carrying out the assessments will be masked to intervention allocated and/or received. Masking will be maintained using a wide range of procedures, including separate offices for the therapists and research assistants carrying out assessments (where they are located in the same building), protocols for answering telephones, message taking and secretarial support, separate diaries, pigeonholes and data file security, and using passwords and encryption of randomisation information.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BeatIt2 for depression alongside Treatment as usual (TAU) (Experimental): BeatIt2 treatment manual and materials are developed and modelled for people with severe/profound learning disabilities. They are designed to be delivered to the person alongside a family or paid carer providing them with regular support, on an outreach basis. It is a structured, time limited, manualised psychological therapy, developed to treat those with learning disabilities and depressive symptoms.
  There is an initial training session for carers regarding their role in the treatment, then 12 sessions with the person with a learning disability and their carer, held weekly or fortnightly, spanning approximately 6 months.
  Activities are carried out with the individuals with learning disabilities at each session and elements of the intervention are delivered via carers. The three main phases are: i) assessment and socialisation into the intervention and establishing a relationship with the person with the disability, ii) working towards change, and iii) finishing therapy.
  Interventions: Behavioral: Behavioural Activation for depression (BeatIt2)
- Treatment as usual (No Intervention): This will include the existing treatments available in NHS and social care for adults with learning disability with depression, including anti-depressants, mood stabilizers, and any available nursing and psychological supports/interventions. Additionally, for all those in the study, the investigators will provide their General Practitioner and specialist services with a summary of the NICE guidelines on treatment of depression for adults with learning disabilities.

INTERVENTIONS:
Behavioral: Behavioural Activation for depression (BeatIt2) — It is a structured, time limited, manualised psychological therapy, developed to treat those with learning disabilities and depressive symptoms.
  There is an initial training session for carers regarding their role in the treatment, then 12 sessions with the person with a learning disability and their carer, held weekly or fortnightly, spanning approximately 6 months.
  Activities are carried out with the individuals with learning disabilities at each session and elements of the intervention are delivered via carers. The three main phases are: i) assessment and socialisation into the intervention and establishing a relationship with the person with the disability, ii) working towards change, and iii) finishing therapy. The first phase includes assessment of the person's pattern of daily activity, barriers and facilitators to engaging in activity, and examining the link between activity and mood. Specific attention is given to the role of communication and how scaffolding can be provid
  Arms: BeatIt2 for depression alongside Treatment as usual (TAU)

SUMMARY:
Research shows that people with severe learning disabilities get depressed at least as often as the wider population. Psychological therapies are recommended to treat depression, and some of these have been adapted for those people with learning disabilities who can talk about their problems. No research has properly tested a psychological therapy for people with severe learning disabilities and any mental health problem. The investigators recently completed a study that tested a psychological therapy (behavioural activation) for people with mild learning disabilities and depression. Behavioural activation improves people's mood by helping them to re-engage in activity that has meaning and purpose for them, rather than relying on talking or thinking skills. Because of this behavioural activation might be promising for people with severe learning disabilities and depression. Along with PAMIS, an organisation for families of people with more profound disabilities, the investigators have adapted the therapy for this group. The investigators now want to find out if it would be possible to carry out a research project about whether behavioural activation works for depressed adults with severe learning disabilities. This is called a feasibility study. The investigators would see if it is possible to recruit 50 adults with severe learning disabilities, and if they are willing to be randomly placed in a group who get behavioural activation or a group who get usual help from services. Other information about running a study would be collected, including about keeping in contact with participants and what measures are needed to find out if change is happening.

DETAILED DESCRIPTION:
People with severe and profound learning disabilities have significant lifelong impairment of general intelligence (IQ<40 with associated adaptive skill deficits). They have high support needs and limited or no verbal communication.

Prevalence of depression is increasing for people with learning disabilities (from 12.6% in 2016/17 to 14.5% in 2021/22 in England). The main treatment in use is medication, and antidepressant use is rising.

The 2016 NICE guideline on mental health problems in people with learning disabilities found the only available evidence on psychological interventions for depression was very low quality for specially adapted Cognitive Behavioural Therapy (CBT), and only for people with mild/moderate learning disabilities. Only three RCTs (total n=130) and three controlled before-and-after studies (total n=130) of CBT were identified for all mental health conditions. There was no evidence for people with severe learning disabilities, and CBT is not accessible to people with significant communication and cognitive limitations. The NICE included research recommendations for psychosocial intervention RCTs for people with severe learning disabilities and mental health problems.

Behavioural Activation (BA) uses behavioural principles to treat depression and is probably more accessible to people with severe learning disabilities than wholly talking therapies like CBT. The core aims of BA are: i) to reduce general avoidance of activity, commonly associated with depression, and ii) to increase engagement in valued and purposeful activity. In the general population, BA is at least as effective as antidepressant medications and superior or non-inferior to CBT, pill-placebo, and treatment as usual; and has effects as lasting as CBT following treatment termination.

The investigators aim to examine the feasibility of completing a two arm RCT of an adapted version of behavioural activation for people with severe to profound intellectual disabilities (BeatIt2), with participants randomised to BeatIt2 alongside treatment as usual (TAU) or to TAU alone.

Research questions concern: i) recruitment, ii) retention 12 months post-randomisation, iii) outcome measures with greatest utility in detecting meaningful change, and iv) whether adverse events occur.

A process evaluation will also be carried out, bringing together evidence on: v) acceptability of the intervention across families, paid carers and services, vi) fidelity of therapy delivery and adherence to the manual, vii) feasibility of collecting service use and quality of life data from adults with severe learning disabilities from both arms of the study (to test the feasibility of a later health economic study), and viii) the mechanisms of change and how the context of the intervention affects implementation.

ELIGIBILITY:
Inclusion Criteria:

* Administratively defined severe/profound learning disabilities, confirmed by carer report using the Vineland Adaptive Behaviour Scales 3rd edition. A severe/profound learning disability will be confirmed by an ABC composite score of 50 or below (Sparrow et al., 2016). Individuals with severe/profound learning disabilities can be characterised by high support needs, limited or no expressive or receptive verbal communication, and significant impairments across adaptive functioning skills.
* 18 years old and over
* Clinically significant unipolar depression, meeting the Diagnostic Criteria for Psychiatric Disorders for use with Adults with Learning Disabilities
* Has a family member or paid carer who has supported them for a minimum of 6 months to complete the screening and baseline visits OR is able to obtain information for the previous 4 months prior to randomisation. The carer, or another named individual, should be available for weekly-fortnightly treatment sessions with the practitioner, and should currently provide a minimum of 10 hours support per week to the participant.

Exclusion Criteria:

* Mild/moderate learning disabilities
* A presentation judged by the research team as likely to interfere with the successful engagement with the intervention (e.g. severe agitation, late-stage dementia, uncontrolled epilepsy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-04 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Intellectual Disabilities Depression Scale (IDDS) | Baseline, 4, 6, 8, 12 months post-baseline
  This is a 38-item behavioural checklist derived from DSM-III-R criteria, designed to measure the frequency of identified depressive behaviours within a four-week period. Minimum possible score is 0 and maximum possible score is 228. Higher scores indicate a higher frequency of depressive symptoms.

SECONDARY OUTCOMES:
Anxiety Depression and Mood Scale (ADAMS) | Baseline & 12 months post-baseline
  This scale is the only one that has been shown to be a reliable and valid measure of anxiety in adults with severe/profound intellectual disabilities. Since the investigators are already using two measures of depressive symptoms, only the anxiety sub-scale of the Anxiety, Depression and Mood Scale will be used in this study. Seven items will be used from the original 28-item measure. These items comprise the 'generalised anxiety' subscale, with informants reporting on their observations of these symptoms in the last 2 weeks. Items are scored on a four-point Likert scale that combines frequency and severity of symptoms. Minimum possible score is 0 and maximum possible score is 42. Higher scores indicate a higher frequency and severity of anxiety symptoms.
Index of Community Involvement | Baseline & 12 months post-baseline
  This 16-item scale provides a measure of participation in social and community based activities during the previous 4 weeks. Minimum possible score is 0 and maximum is 80. Higher scores indicate a higher frequency of engagement in community activities.
Index of Participation in Domestic Life | Baseline & 12 months post-baseline
  This scale measures participation in 13 household tasks during the previous 4 weeks. Minimum possible score is 0 and maximum possible score is 26. Higher scores indicate higher levels of independent participation in domestic tasks.
EQ-5D-5L | Baseline & 12 months post-baseline
  This proxy report questionnaire assesses the participants' health related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has five levels: no problems, slight problems, moderate problems, severe problems and extreme problems. Possible minimum score is 5 and possible maximum score is 25. Higher scores indicate more problems in these domains. There is an additional visual analogue scale with endpoints of 'the worst health you can image' and 'the best health you can image' on a 0 to 100 scale.
The Behaviour Problems Inventory - Short form (BPI-S) | Baseline & 12 months post-baseline
  The BPI-S is an informant-based behaviour rating instrument for adults with intellectual disabilities who display challenging behaviour. It is a 30-item measure which includes three subscales: Self-Injurious Behaviour (14 items), Stereotyped Behaviour (24 items), and Aggressive/Destructive Behaviour (11 items). This measure assesses both severity and frequency. The frequency of the BPI-S measure is rated on a 5-point Likert scale ranging from 0 (never/no problem) to 4 (hourly). The severity of the self-injurious and aggressive/destructive behaviour is rated on a 3-point Likert scale starting from 1 (mild) to 3 (severe). Possible minimum and maximum scores are 0 - 56 (self-injurious behaviours), 0 - 70 (aggressive/destructive behaviours), and 0 - 48 (stereotyped behaviours). Higher scores indicate a higher frequency and severity of problem behaviours.
Emotional Difficulties Self-Efficacy Scale | Baseline & 12 months post-baseline
  This is a flexible five item scale to assess carer (parents and paid carer) perceptions of their self-efficacy in specific support domains relating to children and adults with intellectual disability or autism. Minimum possible score is 0 and maximum possible score is 80. Higher scores indicate higher perceived self-efficacy.
Warwick Edinburgh Mental Wellbeing Scale | Baseline & 12 months post-baseline
  This seven item self-report measure of mental wellbeing has strong internal consistency (Cronbach's alpha = 0.88 - 0.93) and has proven to have good construct validity, with significant correlations with scores from other standardised measures of mental health and wellbeing, the PHQ-9 and GAD-7. The possible minimum score is 13 and possible maximum score is 65. Higher scores indicate higher levels of wellbeing.
Client Service Receipt Inventory (CSRI) | Baseline, 4, 6, 8, 12 months post-baseline
  CSRI is a validated tool to measure total package resource use and has been used in evaluations involving people with learning disabilities. It records items such as contacts with community-based primary care, other health or social services, educational services, and outpatient and inpatient attendances. Unit costs for most of these are available.
Medication Inventory | Baseline, 4, 6, 8, 12 months post-baseline
  Medication use will be recorded, and any changes in use of medication over the course of the intervention and during follow-up will be noted to determine if there are treatment differences between the two arms of the study. In combination with the CSRI, medication use will also be costed.
The Mood Interest and Pleasure Questionnaire | Baseline and 12-months post-baseline
  This comprises 12 items from two subscales (mood, and interest and pleasure) and requires proxy respondents to indicate how often a particular symptom has occurred within the last 2 weeks. Possible minimum and maximum scores for each sub-scale are 0 - 24. Lower scores indicate lower mood and lower levels of interest and pleasure. The mood interest and pleasure questionnaire (Ross et al., 2008; Ross & Oliver, 2003) short form shows high internal con sistency (Cronbach alpha coefficients: total = .88; mood = .79; inter est and pleasure = .87) (Ross et al., 2008)